CLINICAL TRIAL: NCT04405180
Title: Nitrites, Skeletal Muscle Mitochondrial Bioenergetics, and Physical Activity in Old Age
Acronym: Nitrite
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gladwin, Mark, MD (Individual)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Daniel Forman, MD, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY20110334; R01AG058883 (NIH)
Record Dates: First submitted 2019-04-15; First posted 2020-05-28 (Actual); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Aging; Sedentary Lifestyle; Frailty
Keywords: 70 and Older; Bioenergetics; Frailty
MeSH Terms: conditions — Sedentary Behavior; Frailty

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple: Participant, Care Provider, Investigator, Outcome Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- 20 mg Sodium Nitrite TID Arm (Experimental): Subject is to receive active study drug three times per day during treatment (12 weeks +/- 5 days) period and then after the treatment period (up to 16 weeks total).
  Interventions: Drug: 20mg sodium nitrite tid
- Placebo Control Arm (Placebo Comparator): Subject is to receive placebo three times per day during treatment period (12 weeks +/- 5 days) and then after the treatment testing period (up to 16 weeks total).
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Placebos — Oral placebo capsule at a dose of 20 mg administered three times per day, during the day.
  Other Names: Placebo
  Arms: Placebo Control Arm
Drug: 20mg sodium nitrite tid — Oral, inorganic sodium nitrite capsule at a dose of 20 mg administered three times per day, during the day.
  Arms: 20 mg Sodium Nitrite TID Arm

SUMMARY:
This 2-site randomized double blinded controlled trial is to confirm and more definitively clarify the impact of a 12-week course of nitrite versus placebo on mitochondrial bioenergetics in older sedentary adults. This investigator will take an integrative physiology approach to determine the effect of nitrite therapy on a comprehensive assessment of mitochondrial energetics, skeletal muscle vascular function, and whole body physical function (cardiorespiratory function, exercise endurance, strength, balance, and physical activity) and fatigability.

DETAILED DESCRIPTION:
Old age is associated with declining skeletal muscle mitochondrial bioenergetics with related decrements in cardiorespiratory fitness (CRF) and physical function that predispose to frailty, disability, and diminished quality of life. While exercise training may moderate and possibly even reverse declines in mitochondrial bioenergetics, potential for such benefit is typically confounded by exercise intolerance with early fatigability that results from the same age-related mitochondrial declines. Consequently, sedentariness is endemic and insidious among the growing population of older adults. This trial is to study the utility of inorganic nitrite salts as a novel means to modify this detrimental pattern. Classic studies demonstrate that nitrite facilitates hypoxic vasodilation in muscle. This investigator's preliminary data suggests that nitrite treatment also augments skeletal muscle mitochondrial bioenergetics in older adults. This investigator proposes improving mitochondrial function will also be reflected in clinical parameters, including CRF as well as broader functional attributes (endurance, strength, and balance) that enable physical activity (PA) and opportunity to mitigate frailty and disability. As such, this application is in line with the National Institute on Aging's mission to develop targeted interventions to prevent and treat age-associated conditions. This multi-disciplinary team has published seminal work indicating that mitochondrial bioenergetics and CRF are significant determinants of physical function in older adults. In parallel efforts, this investigative team showed efficacy of chronic nitrite therapy to improve mitochondrial bioenergetics in older sedentary adults. Only one month of nitrite therapy significantly improved ex vivo assessments of mitochondrial energetics in skeletal muscle biopsies, concomitant with increased skeletal muscle sirtuin-3 expression, a nicotinamide adenine dinucleotide (NAD) dependent lysine deacetylase and key regulator of mitochondrial metabolism. These key data reinforce the premise that nitrite enhances vital mitochondrial metabolism in older adults. Moreover, improvement in muscle energetics in nitrite-treated older adults was linked with increased exercise efficiency as evidenced by reduced oxygen consumption (VO2) during submaximal steady-state walking. This data supports the hypothesis that nitrite will make physical function easier such that physical activity will increase.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years
* Sedentary (<1 hour/week of volitional exercise activity)
* Clinically stable (euvolemic; baseline HR <100 bpm) and without hospitalization or invasive cardiac procedure for 6 weeks

Exclusion Criteria:

* Blood pressure <110 or >160/95 mmHg
* Orthopedic or other chronic condition which limits physical activity or exercise testing assessments
* If valve replacement has been performed, patient may not be enrolled for 12 months after this procedure
* Severe peripheral or pulmonary artery disease
* Anemia: Hgb <11.0 (♂),10.0 (♀) gm/dl
* Participants with diabetes whose HgbA1c >10.0%
* Chronic alcohol (>14 drinks ETOH a week) or drug (any cocaine, methamphetamine, and cannabis ≥4 x week) dependency
* Allergy to lidocaine and red dye
* Chronic use of oral corticosteroids or other medications that affect muscle function
* Current use of organic nitrates or phosphodiesterase type 5 (PDE5) inhibitors
* Unable to hold warfarin, direct-acting oral anticoagulants (DOACs), non-steroidal anti-inflammatory medications (NSAIDs) or aspirin for 3 days prior to muscle biopsy, or to hold thienopyridine medications for 5 days prior to muscle biopsy. Participants unable or unwilling to hold will follow the modified ASA hold plan
* Any bleeding disorder that would contraindicate biopsy such as history of clinically significant bleeding diathesis (e.g., Hemophilia A or B, Von Willebrand's Disease or congenital Factor VII deficiency)
* Unstable psychiatric diagnosis that would affect adherence and ability to complete the protocol
* Dementia or inability to give informed consent or follow study protocol
* End-stage disease
* Other chronic unstable disease such as active neoplasm, end stage chronic kidney, liver or other organ disease

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-04-23 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-07-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University Of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
De-Identified data may be shared with other future investigators as research questions arise.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: A limit in time frame of sharing has not been defined.
Access Criteria: Only de-identified data approved for sharing by PI.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 20 mg Sodium Nitrite TID Arm | Placebo Control Arm
Started | 32 | 32
Completed | 32 | 32
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 20 mg Sodium Nitrite TID Arm | Placebo Control Arm | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.3 (5.4) | 76.1 (6.0) | 75.7 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 28
  Male | 17 | 19 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 32 | 31 | 63
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 1 | 6
  White | 27 | 30 | 57
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Skeletal Muscle Mitochondrial Respiration State 3; Baseline to 12-week Change.
Description: High resolution respirometry via Oroboros Oxygraph 2k is used to assess the effects of 12 weeks of inorganic nitrite vs placebo on skeletal muscle mitochondrial respiration from samples obtained via vastus lateralis muscle biopsy.
Time Frame: 12-week course of study drug supplementation, up to 16 weeks total
Measure: Mean (Standard Deviation); unit: pmol O2/s/mg DW
Arm/Group | 20 mg Sodium Nitrite TID Arm | Placebo Control Arm
Number analyzed (Participants) | 32 | 32
pmol O2/s/mg DW | 2.2 (23.4) | -0.8 (18.4)
Statistical Analysis 1: Comparison: 20 mg Sodium Nitrite TID Arm vs Placebo Control Arm; Test type: Superiority; p = 0.9017, ANCOVA — Adjusted for baseline value of outcome as a covariate using general linear (mixed) models and with multiple imputation for missing data; Mean Difference (Net) = 0.5, Standard Error of Mean 4.0

2. Secondary Outcome: Skeletal Muscle Adenosine Triphosphate (ATP) Production, Baseline to 12-week Change
Description: Using phosphorus-magnetic resonance spectroscopy, we will measure ATPmax (recovery rate) and how it will change after 12 weeks (up to 16 weeks) of inorganic nitrite supplementation vs placebo
Time Frame: 12-week course of study drug supplementation, up to 16 weeks total
Measure: Mean (Standard Deviation); unit: mM ATP/s
Arm/Group | 20 mg Sodium Nitrite TID Arm | Placebo Control Arm
Number analyzed (Participants) | 12 | 13
mM ATP/s | 0.0222 (0.1223) | -0.0131 (0.1263)
Statistical Analysis 1: Comparison: 20 mg Sodium Nitrite TID Arm vs Placebo Control Arm; Adjusted for baseline value of outcome as a covariate using general linear (mixed) models and with multiple imputation for missing data; Test type: Superiority; p = 0.4215, ANCOVA; Mean Difference (Net) = 0.0342, Standard Error of Mean 0.0417

3. Other Pre Specified Outcome: Cardiorespiratory Fitness Measured as Peak Oxygen Uptake (Non-weight Normalized VO2) During a Progressive Resistance Cycle Ergometer Exercise Test; Baseline to 12-week Change
Description: Cardiorespiratory fitness is measured as peak oxygen utilization (non-weight normalized VO2) during a progressive resistance cycle ergometer exercise test that is symptom-limited (maximum).
  This is assessed before and after 12 weeks (16 weeks total) of oral inorganic nitrite supplementation vs placebo.
Time Frame: 12-week course of study drug supplementation, up to 16 weeks total
Measure: Mean (Standard Deviation); unit: ml/minute
Arm/Group | 20 mg Sodium Nitrite TID Arm | Placebo Control Arm
Number analyzed (Participants) | 32 | 32
ml/minute | -50 (212) | -82 (192)
Statistical Analysis 1: Comparison: 20 mg Sodium Nitrite TID Arm vs Placebo Control Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = .9024, ANCOVA; Mean Difference (Net) = 6, Standard Error of Mean 53

4. Other Pre Specified Outcome: Oxygen Utilization (Non-weight Normalized VO2) During a Slow (1.5 Mph) Fixed Rate Walking Speed Test; Baseline to 12-week Change
Description: Oxygen utilization (non-weight normalized VO2) is measured during slow walking during the last minute of a 5-minute slow (1.5 mph) fixed rate walking speed test.
  This is assessed before and after 12 weeks (16 weeks total) of oral inorganic nitrite supplementation vs placebo.
Time Frame: 12-week course of study drug supplementation, up to 16 weeks total
Measure: Mean (Standard Deviation); unit: ml/minute
Arm/Group | 20 mg Sodium Nitrite TID Arm | Placebo Control Arm
Number analyzed (Participants) | 32 | 32
ml/minute | -92 (123) | -35 (188)
Statistical Analysis 1: Comparison: 20 mg Sodium Nitrite TID Arm vs Placebo Control Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.1646, Mixed Models Analysis; Mean Difference (Net) = -59, Standard Error of Mean 42

5. Other Pre Specified Outcome: Endurance During a Submaximal Constant Workload Cycle Ergometer Exercise Test; Baseline to 12-week Change.
Description: Endurance is measured as duration (minutes) of exercise during a constant submaximal workload cycle ergometer exercise (i.e., calibrated at 75-80% of the maximum resistance [watts] achieved in a prior maximum cycle ergometer exercise test).
  This is assessed before and after 12 weeks (16 weeks total) of oral inorganic nitrite supplementation vs placebo.
Time Frame: 12-week course of study drug supplementation, up to 16 weeks total
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 20 mg Sodium Nitrite TID Arm | Placebo Control Arm
Number analyzed (Participants) | 32 | 32
minutes | 0.8 (3.8) | -0.1 (4.5)
Statistical Analysis 1: Comparison: 20 mg Sodium Nitrite TID Arm vs Placebo Control Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.9814, ANCOVA; Mean Difference (Net) = 0.0, Standard Error of Mean 1.2

6. Other Pre Specified Outcome: Time to Complete a Fast-paced 400 m Corridor Walk; Baseline to 12-week Change
Description: Time to complete a fast-paced 400 m corridor walk is assessed
  This is assessed before and after 12 weeks (16 weeks total) of oral inorganic nitrite supplementation vs placebo.
Time Frame: 12-week course of study drug supplementation, up to 16 weeks total
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | 20 mg Sodium Nitrite TID Arm | Placebo Control Arm
Number analyzed (Participants) | 32 | 32
minutes | 0.0 (0.9) | -0.2 (0.9)
Statistical Analysis 1: Comparison: 20 mg Sodium Nitrite TID Arm vs Placebo Control Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.6217, Mixed Models Analysis; Mean Difference (Net) = 0.1, Standard Error of Mean 0.3

7. Other Pre Specified Outcome: Borg Rating of Perceived Exertion During a 5-minute Slow (1.5 Mph) Fixed Rate Walking Speed Test; Baseline to 12-week Change
Description: Fatigability is assessed using the Borg Rating of Perceived Exertion during minute 5 of a 5-minute fixed rate (1.5 mph) slow walking test. Borg Rating of Perceived Exertion is scored on a scale from 6 to 20 with 6 being the least difficult or intense (better) and 20 being the most difficult or intense (worse).
  This is assessed before and after 12 weeks (up to 16-weeks) of inorganic nitrite supplementation vs placebo.
Time Frame: 12-week course of study drug supplementation, up to 16 weeks total
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 20 mg Sodium Nitrite TID Arm | Placebo Control Arm
Number analyzed (Participants) | 32 | 32
score on a scale | -0.3 (1.4) | -0.5 (2.2)
Statistical Analysis 1: Comparison: 20 mg Sodium Nitrite TID Arm vs Placebo Control Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.7981, Mixed Models Analysis; Mean Difference (Net) = -0.1, Standard Error of Mean 0.5

8. Other Pre Specified Outcome: Short Physical Performance Battery; Baseline to 12-week Change
Description: The Short Physical Performance Battery is assessed before and after 12-weeks (up to 16-weeks) of inorganic nitrite supplementation vs placebo. The Short Physical Performance Battery score is the aggregate of three sub-scales for balance, gait speed and repeated sit to stand performance. Each of the three sub-scales is scored from 0 to 4 with 0 being the poorest performance and 4 being the best performance. The scores for balance, gait speed, and repeated sit to stand performance are add for a total score ranging from 0 (worst) to 12 (best).
Time Frame: 12-week course of study drug supplementation, up to 16 weeks total
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 20 mg Sodium Nitrite TID Arm | Placebo Control Arm
Number analyzed (Participants) | 32 | 32
score on a scale | -0.1 (1.9) | 0.4 (1.5)
Statistical Analysis 1: Comparison: 20 mg Sodium Nitrite TID Arm vs Placebo Control Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.6677, Mixed Models Analysis; Mean Difference (Net) = -0.2, Standard Error of Mean 0.4

9. Other Pre Specified Outcome: Grip Strength; Baseline to 12-week Change
Description: Maximum grip strength is assessed before and after 12 weeks (up to 16-weeks) of inorganic nitrite supplementation vs placebo.
Time Frame: 12-week course of study drug supplementation, up to 16 weeks total
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | 20 mg Sodium Nitrite TID Arm | Placebo Control Arm
Number analyzed (Participants) | 32 | 32
kg | 1.3 (3.8) | -0.5 (2.9)
Statistical Analysis 1: Comparison: 20 mg Sodium Nitrite TID Arm vs Placebo Control Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.3745, Mixed Models Analysis; Mean Difference (Net) = 1.0, Standard Error of Mean 1.1

10. Other Pre Specified Outcome: Physical Activity (Accelerometry), Measured as Daily Step Count; Baseline to 12-week Change
Description: Physical activity is measured as daily step count (assessed using an Actigraph accelerometry device on the participant's wrist), before and after 12 weeks (up to 16-weeks) of inorganic nitrite supplementation vs placebo.
Time Frame: 12-week course of study drug supplementation, up to 16 weeks total
Measure: Mean (Standard Deviation); unit: steps
Arm/Group | 20 mg Sodium Nitrite TID Arm | Placebo Control Arm
Number analyzed (Participants) | 32 | 32
steps | 118 (1244) | -180 (954)
Statistical Analysis 1: Comparison: 20 mg Sodium Nitrite TID Arm vs Placebo Control Arm; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.5496, ANCOVA; Mean Difference (Net) = 243, Standard Error of Mean 400

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | 20 mg Sodium Nitrite TID Arm | Placebo Control Arm
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 1/32
Other Adverse Events (participants affected / at risk) | 10/32 | 14/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 mg Sodium Nitrite TID Arm (N=32) | Placebo Control Arm (N=32)
Other (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20 mg Sodium Nitrite TID Arm (N=32) | Placebo Control Arm (N=32)
Gastroesophogeal Reflux Disease (Gastrointestinal disorders) | 1 | 0
(Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Upper Respiratory Infection (Infections and infestations) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 0 | 2
Other (Infections and infestations) | 3 | 6
Fall (Injury, poisoning and procedural complications) | 1 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 1
Urinary Tract Pain (Renal and urinary disorders) | 0 | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Departures from the muscle preservation protocol resulted in widespread ice artifact in the majority of mounted tissue samples. Nearly all muscle samples are non-viable for histological and morphological analyses. Consequently, skeletal muscle histological and morphological outcomes (cross sectional area, fiber type, fiber type area, and mitochondrial content) were omitted due to to technical limitations and predominant doubts regarding the reliability of the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT04405180/Prot_SAP_002.pdf
  • Informed Consent Form (2024-09-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT04405180/ICF_003.pdf